CLINICAL TRIAL: NCT07158411
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Effect of Vimseltinib on Organic Cation Transporter 2 (OCT2) Inhibition in Healthy Male Participants
Brief Title: Evaluate the Effect of Vimseltinib on Organic Cation Transporter 2 (OCT2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: DCC-3014-01-008
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metformin + Vimseltinib (Experimental): Metformin as single dose will be administered on Day 1 and Day 6. Vimseltinib will be administered every day (QD) on Days 3 through 6
  Interventions: Drug: Vimseltinib; Drug: Metformin

INTERVENTIONS:
Drug: Vimseltinib — Administered orally
Drug: Metformin — Administered orally

SUMMARY:
The main purpose of this study is to evaluate the effect of multiple doses of vimseltinib on the pharmacokinetics (PK) of a clinical OCT2 substrate (metformin) in healthy male participants. This study will also assess the safety and tolerability when vimseltinib is co-administered with the clinical OCT2 substrate (metformin) in healthy male participants. This study will last approximately 25 days.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) from 18 to 32 kilogram per square meter (kg/m^2).
2. Participants are in good general health, as required by the protocol and as determined by Principal Investigator.
3. Adequate organ function and blood and urine tests, as required by the protocol and as determined by Principal Investigator.

Exclusion Criteria:

1. History or presence of clinically significant diseases of the neurological, dermatological, renal, hepatic, gastrointestinal, cardiovascular, or musculoskeletal systems and/or history or presence of clinically significant psychiatric, immunological, endocrine, or metabolic disease in the opinion of the Investigator.
2. Unwilling or unable to comply with the requirements of the protocol.
3. Determined by Principal Investigator to be unsuitable to participate in the study for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 22 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK): Maximum Observed Plasma Drug Concentration (Cmax) of Metformin | Predose up to 48 hours postdose
PK: Area Under the Concentration Versus Time Curve (AUC) of Metformin | Predose up to 48 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline through Day 25

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No